CLINICAL TRIAL: NCT06070415
Title: Adherence to Home Treatment of Patients With Low Back Pain Through the Use of Information and Communication Technologies.
Brief Title: Adherence to Exercises for Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, University teacher, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHATBOT_LOW_BACK_PAIN
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Treatment Adherence; Treatment Compliance
Keywords: Treatment adherence; New technologies; Lowback pain
MeSH Terms: conditions — Treatment Adherence and Compliance; Patient Compliance | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two arms study, experimental vs control
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The interventor providing the education sessions will be blinded to group allocation The outcome assessor will be blinded to the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Home exercise assisted with a chatbot
  Interventions: Device: Chatbot; Other: Education
- Control (Active Comparator): Home exercise, usual care
  Interventions: Other: Home exercise, usual care; Other: Education

INTERVENTIONS:
Device: Chatbot — 12 week- intervention consisting of messages with an explanatory video of each exercise indicating how to do it and how many repetitions to perform
  Arms: Experimental
Other: Home exercise, usual care — 12 week- intervention. Printed sheets indicating how to exercises and how many repetitions to perform
  Arms: Control
Other: Education — One-week, three sessions in alternate days, outpatient supervised education on how to perform the exercises at home

SUMMARY:
This project focuses on the effectiveness of a Chatbot in promoting adherence to home physiotherapy treatment for patients with lumbar musculoskeletal injuries. The use of digital technologies and media are an important option to complement in-person treatment and promote adherence to treatment at home. The research aims to verify whether the use of a Chatbot as a means of communication can produce improvements in patient adherence and clinical results.

DETAILED DESCRIPTION:
Currently, performing therapeutic exercises in the treatment of musculoskeletal injuries of the spine is decisive in many cases to achieve an improvement in the symptoms of these pathologies, both in the patient's functionality and in the patient's evaluation of their pain. These types of exercises provide improvement, whether they are outpatient or at home. Due to the paradigm shift that has occurred in recent years, mainly motivated by limited resources and the COVID-19 pandemic, it is necessary to complement in-person exercise and/or teaching sessions with homework whenever possible. In addition, unnecessary travel is avoided in case patients live far from the consultation.

Adherence to treatment is crucial to obtain the desired benefits. According to the WHO (2003), adherence is the degree to which a person's behavior corresponds to the recommendations agreed upon by a healthcare professional, and it has been observed that patients who comply may have a better outcome at the end of treatment. However, not meeting a minimum of more than 65% adherence negatively influences the outcome of the patient's recovery, with probable consequences on socio-health costs.

Before the appearance of new technologies, home-type therapeutic exercises were taught in consultation and given to the patient in paper format. Nowadays, the use of information and communication technologies (ICT) and digital media are an option when administering home treatments, and thanks to these we have much more complete teaching materials. when it comes to remembering what was learned in consultation, such as the Chatbot. For this reason, we value the possibility that the use of this system can help increase adherence to treatment and therefore improve your health condition.

On the other hand, non-compliance rates with treatment are one of the main barriers when it comes to obtaining benefits for the patient. Therefore, digital applications in physiotherapy should be aimed at improving clinical outcomes and promoting adherence through interactive and accessible environments that promote self-efficacy and changes in behavior and routines, as offered by the Chatbot program. One of the most common forms of ICT use is through the use of smartphones, where half of the users of these devices use them to obtain information about health issues, and a fifth uses applications related to this area. This has expanded the offer of health-oriented mobile applications but very little research has been carried out to evaluate adherence or the level of satisfaction among users.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Diagnosis of lumbar pain.
* Indication of treatment through home exercises.
* With a personal smartphone
* Verbally confirms to have installed an instant messaging service or app, and accesses it at least 3 times a week

Exclusion Criteria:

* No to sign the informed consent.
* Not able to understand, read and write in the Spanish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Adherence | 0 weeks, 12 weeks
  Record of the number of sessions performed.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 0 weeks, 12 weeks
  Numerical scale from 0 to 10, where 0 indicates no pain and 10 is the maximum pain experienced.
Disability | 0 weeks, 12 weeks
  The Oswetry Disability Index (ODI) scale, each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Satisfaction scale with the treatment received | 12 weeks
  The CRES-4 satisfaction scale consists of four items designed to evaluate whether patients are satisfied with the therapy they have received and whether it has been perceived as effective. Its global score is intended to reflect treatment effectiveness as perceived by the patient. It is a good complementary tool to judge, in particular, satisfaction with the treatment received. Consists of four questions, and score with a score ranging from 0 to 18 points. The more points, the more satisfied you are with the treatment.
Sistem usability scale | 12 weeks
  It consists of a 10 item questionnaire for measuring the usability of the experimental intervention tool with five response options for respondents, from Strongly agree to Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, Principal Investigator — University of Valencia
Locations (1):
- David Hernández Guillén, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No